CLINICAL TRIAL: NCT00005786
Title: A Pilot Study of Arsenic Trioxide in the Treatment of Relapsed and Refractory Indolent Lymphomas
Brief Title: Arsenic Trioxide in Treating Patients With Relapsed or Refractory Lymphoma or Leukemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00040; GCO # 99-884 ME*; R01CA085748 (NIH); CDR0000067719 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Prolymphocytic Leukemia; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Leukemia, Prolymphocytic; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Arsenic Trioxide

ARMS (1):
- Treatment (arsenic trioxide) (Experimental): Patients receive arsenic trioxide IV over 1-4 hours on days 1-5. Treatment repeats every 21 days for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression. Patients with responding or stable disease may receive 6 additional courses.
  Interventions: Drug: arsenic trioxide; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: arsenic trioxide — Given IV
  Other Names: Arsenic (III) Oxide; Arsenic Sesquioxide; Arsenous Acid Anhydride; AS2O3; Trisenox
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have relapsed or refractory lymphoma or leukemia. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and toxicity profile of arsenic trioxide in patients with relapsed or refractory low-grade lymphomas.

II. To determine the incidence of complete and partial responses to arsenic trioxide in patients with previously treated low-grade lymphomas.

III. To evaluate basic science correlates of arsenic trioxide activity in order to improve our understanding of the mechanism of action for arsenic trioxide in patients with low-grade lymphomas.

OUTLINE: This is a nonrandomized, open-label study.

Patients receive arsenic trioxide IV over 1-4 hours on days 1-5. Treatment repeats every 21 days for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression. Patients with responding or stable disease may receive 6 additional courses.

Patients are followed every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of relapsed or refractory low-grade lymphoma
* Patients must have disease that has relapsed from or is refractory to standard cytotoxic therapy; patients must have received at least one standard cytotoxic drug regimen; there is no limit on the number of prior therapies, including high dose chemotherapy regimens, provided the patient has recovered from prior toxicities; relapsed disease is defined as the development of lymphadenopathy, splenomegaly, malignant lymphocytosis greater than 5,000, or infiltration of the bone marrow with malignant lymphocytes in a patient who had previously achieved a response of at least six months in duration; refractory disease is defined as never achieving a PR or a CR or PR that is less than six months in duration; prior total body irradiation is not allowed; radiation to individual site is permitted, and is not included as a regimen
* Serum creatinine =< 2.0 mg/dl
* Total bilirubin =< 2.0 mg/dl
* Serum SGOT, SGPT =< 2.5 times the upper limit of institutional normal
* Patients who are female and have childbearing potential must have a negative pregnancy test; all patients who are engaging in sexual intercourse that may result in a pregnancy must use appropriate contraception while receiving treatment on this protocol
* Patients must have sufficient mental capacity to understand the explanation of the study and to give his or her informed signed consent
* Patients must display Karnofsky performance status of 60% or greater
* Patients should have a life expectancy of > 12 weeks so as to permit adequate follow-up of toxicity
* Patients must have recovered from the toxicity of recent therapy prior to enrollment in this study
* Absolute neutrophil count > 1500/uL, unless cytopenias are the result of bone marrow infiltration by lymphoma; permission of the protocol PI is required in this situation
* Platelet count > 75,000/uL, unless cytopenias are the result of bone marrow infiltration by lymphoma; permission of the protocol PI is required in this situation; patients with thrombocytopenia secondary to active ITP or anemia secondary to an active autoimmune hemolytic anemia at the time of evaluation are excluded

Exclusion Criteria:

* Pregnant or lactating women; arsenic compounds could be transferred to the fetus or child with resultant harm
* Concurrent treatment with cytotoxic chemotherapy, radiation or investigational agents; this exclusion does not include concurrent glucocorticoids fro brief durations; patients must have recovered from the toxicity of prior therapy prior to enrollment in this study
* Active serious infections not controlled by antibiotics
* Inability to comply with the treatment protocol or follow-up testing
* Patients with HIV infection; there are currently insufficient data to support the safety of administering arsenic compounds in combination with anti-retroviral drugs
* Patients with active viral or autoimmune hepatitis
* Patients with history of cardiac arrhythmia, heart block, or myocardial infarction within the past 6 months
* Patients with known CNS disease
* Patients requiring amphotericin B therapy
* Patients with significant peripheral neuropathy (>= grade 3), regardless of cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-01; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Toxicity as assessed by Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria version 2.0 | Up to 2 years after completion of study treatment
Incidence of complete and partial response | Up to 2 years

SECONDARY OUTCOMES:
Potential surrogate of arsenic trioxide clinical activity | From baseline to up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Luis Isola, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States